CLINICAL TRIAL: NCT00171639
Title: The Use of Zoledronic Acid in Men on Androgen Deprivation Therapy for Prostate Cancer With Preexisting Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CZOL446EUS72
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: zoledronic acid

SUMMARY:
This study is being conducted to evaluate the effect of an investigational drug on bone loss in men with prostate cancer who are receiving Androgen Deprivation Therapy (ADT).

In order to participate, male patients 18 years and older must be veterans from participating Veterans Administration Medical Centers that are receiving ADT for prostate cancer and have established osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age > 18 years
* Histologically confirmed diagnosis of carcinoma of the prostate
* Stage M0: Patients just starting ADT must be stage M0 [PSA <10 (then bone scan not needed) or negative bone scan (regardless of PSA)]. Patients already on ADT must have been M0 at the initiation of ADT and have maintained a stable, low PSA (< 2.0) on continuous ADT since that time.
* Patients initiating or receiving ADT with a LHRH agonist (with or without an antiandrogen) and with the intended duration of ADT of at least 12 months from the time of randomization. Patients undergoing bilateral orchiectomy or with history of this procedure are also eligible. For patients already on ADT, the therapy must be continuous, and if there is more than one missed or delayed dose (> 1 mo delay) in any one year period, the patient is not eligible.
* Patient with a baseline BMD T-score <-2.0 in the lumbar spine (L2-L4) and/or the total hip are eligible
* Life expectancy of at least 12 months
* Zubrod performance status of 0, 1, or 2

Exclusion Criteria

* Patients who received any bisphosphonate therapy in the past 6 months
* Metabolic bone disease including Paget's disease or hyperparathyroidism or vitamin D deficiency. Patients with vitamin D deficiency or secondary hyperparathyroidism due to vitamin D deficiency may be treated and reassessed for consideration for the trial, as detailed in Appendix 9.
* Radiographic evidence of bone metastases
* Patients who have received treatment with systemic corticosteroids within the past 12 months (short term corticosteroid therapy for up to one month duration, e.g. for acute illness like asthma exacerbation, is acceptable)
* Patients with prior exposure to anabolic steroids or growth hormone within the past 6 months
* Current treatment with estrogen or complementary medicines known to contain estrogens
* Patients with previous or concomitant malignancy within the past 5 years except adequately treated basal or squamous cell carcinoma of the skin, and colonic polyps with non-invasive malignancy which have been removed
* Patients with nonmalignant conditions which would confound the evaluation of the primary endpoint, impair tolerance of therapy, or prevent compliance to the protocol, including:

  * uncontrolled infections
  * uncontrolled type 2 diabetes mellitus
  * diseases with influence on bone metabolism, such as Paget's disease or uncontrolled thyroid or parathyroid dysfunction
  * cardiovascular, renal, hepatic, pulmonary and neurologic/psychiatric diseases which would prevent prolonged follow-up
* Patients with clinical or radiological evidence of existing fracture in the lumbar spine or either hip
* Patients with history of lumbar spine surgery that directly involved the bone or resulted in implanted hardware; or rendered the lumbar spine not evaluable (Some patients with a history of laminectomy alone may qualify).
* Patients with history of unilateral fracture of hip due to trauma or unilateral hip surgery and the other hip and lumbar spine are not evaluable.
* Patients for whom the lumbar spine and at least one hip are not evaluable for any reason.
* Patients treated with systemic investigational drugs(s) and /or device(s) within the past 30 days
* Patients with any prior treatment for osteoporosis except for calcium and vitamin D
* Patients with abnormal renal function as evidenced by either a serum creatinine greater than 3 mg/dL or by a calculated creatinine clearance of 40 ml/minute or less (Use Cockcroft-Gault equation. See Appendix 5).
* Corrected (adjusted for serum albumin) serum calcium concentration < 8.0 mg/dl (2.00 mmol/L)\

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-06; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Percent change in bone mineral density of the lumbar spine (L2-L4) at 6 and 12 months. | 12 months

SECONDARY OUTCOMES:
Percent change in bone mineral density of the total hip (including femoral neck, trochanteric region, and Ward's triangle) following one year of therapy. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nirmala Bhoopalam, MD, Principal Investigator — Hines VA Medical Center
Locations (7):
- United States (7):
  - Southern AZ VA Health Care System, Tucson, Arizona
  - VA Medical Center-Long Beach, Long Beach, California
  - Washington VA Medical Center, Washington D.C., District of Columbia
  - West Side VMAC, Chicago, Illinois
  - Hines VA Medical Center, Hines, Illinois
  - Kansas City VMAC, Kansas City, Missouri
  - VAWNY Buffalo, Buffalo, New York

REFERENCES:
- [Result] Campbell SC, Bhoopalam N, Moritz TE, Pandya M, Iyer P, Vanveldhuizen P, Ellis NK, Thottapurathu L, Garewal H, Warren SR, Friedman N, Reda DJ. The use of zoledronic acid in men receiving androgen deprivation therapy for prostate cancer with severe osteopenia or osteoporosis. Urology. 2010 May;75(5):1138-43. doi: 10.1016/j.urology.2009.11.083. Epub 2010 Mar 19. PMID 20303574